CLINICAL TRIAL: NCT00198458
Title: Clinical Evaluation of Hypersensitivity Reaction to Vitrase (Ovine Hyaluronidase, 150 USP Units/mL) Open Label, Normal Volunteer Study
Brief Title: Hypersensitivity Reaction to Vitrase (Ovine Hyaluronidase)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ISTA-VIT-CS05
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Drug Hypersensitivity
MeSH Terms: conditions — Drug Hypersensitivity | interventions — Chondroitinases and Chondroitin Lyases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrase (Experimental): A single intradermal dose of 4.5 USP units of Vitrase at one site and the same volume of saline at a distant site for comparative control.
  Interventions: Drug: Vitrase

INTERVENTIONS:
Drug: Vitrase
  Other Names: ovine hyaluronidase

SUMMARY:
The objective of this study was to rule out a greater than 10% incidence of hypersensitivity to Vitrase following a single intradermal injection of 3 USP units Vitrase. Less than or equal to a 10% hypersensitivity response was considered acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to avoid disallowed meds

Exclusion Criteria:

* Known hypersensitivity to hyaluronidase and/or bee sting
* Previous known exposure to ovine hyaluronidase or bovine hyaluronidase
* Atopic individuals assessed by medical history
* Topical/inhaled/systemic corticosteroids within 30 days
* Concurrent use of antihistamines or anti-inflammatory during study
* Active or chronic disease likely to affect immune function
* History of alcohol/drug abuse within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2004-07; Primary Completion 2004-07 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity | 1-2 days
  Incidence of hypersensitivity to Vitrase following a single intradermal injection of 4.5 USP units Vitrase.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Grillone, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- Solano Clinical Research (A Division of Dow Pharmaceutical Sciences), Davis, California, United States